CLINICAL TRIAL: NCT06224478
Title: Assessment of Palatal Mucosal Thickness in Different Vertical Skeletal Pattern: a 3D Analysis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, VANDE VANNET Bart, Head of the University Department of Dentofacial Orthopedics, University of Lorraine, Nancy, Central Hospital, Nancy, France
Other Study IDs: 2023PI218
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Palatal Mucosa Thickness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hypodivergent
  Interventions: Other: Measurement of palatal mucosa thickness on CBCT scans
- Normodivergent
  Interventions: Other: Measurement of palatal mucosa thickness on CBCT scans
- Hyperdivergent
  Interventions: Other: Measurement of palatal mucosa thickness on CBCT scans

INTERVENTIONS:
Other: Measurement of palatal mucosa thickness on CBCT scans — Measurement of palatal mucosa thickness on CBCT scans in hypodovergent, normodivergent and hyperdivergent patients

SUMMARY:
This study assesses the potential statistical correlation between vertical facial pattern and palatal mucosa thickness.

Data collection : dicom files (CBCT) merged with STL files of n patients for soft tissue visualization

Aim: to volumetrically assess (with CBCT) the palatal mucosa thickness in different vertical facial types to aid clinicians in the planning and placement of orthodontic miniscrews.

Hypothesis : There is no significant difference between the 3 groups studied (i.e. no correlation between palatal mucosa thickness and vertical facial typology).

DETAILED DESCRIPTION:
Study rationale : The use of palatal miniscrew offers the possibility to improve the effectiveness of orthodontic expansion devices. Palatal expanders supported by miniscrew can be applied with different clinical protocols. The palatal mucosa thickness affects the choice of miniscrew length.

Justification for overlaying on STL files: When the lingual dorsum and palatal mucosa are in mutual contact during CBCT examination, it is not possible to distinguish one from the other during subsequent imaging evaluation. Various methods have been proposed to overcome these limitations, including the superimposition of the dicom and stl files: this methodology enables the profile of the palatal mucosa to be distinctly identified in all the analyzed scans.

ELIGIBILITY:
Inclusion Criteria:

* Full permanent dentition (except for third molar)
* Normal craniofacial development
* Aged > 16 years
* Complete skeletal maturity (assessed by the cervical vertebral maturation method)
* Absence of previous orthodontic or orthognatic surgical treatment

Exclusion Criteria:

* Absence of any tooth other than the third molar
* Maxillary impacted tooth
* CBCT scans taken without teeth in occlusion/open bite
* Distorting pathologies of the facial mass affecting the palatal zone
* Periodontal or endodontic diseases affecting the bone
* Presence of metallic artifact
* History of previous orthognatic or orthodontic surgeries

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have undergone CBCT at Nancy University Hospital, Boston University and in private practice
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-25 (Estimated); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Palatal mucosa thickness | Baseline
  In milimetres